CLINICAL TRIAL: NCT04147728
Title: Stereotactic Radiosurgery Combination With Anlotinib for Limited Brain Metastases With Perilesional Edema in Non-small Cell Lung Cancer：An Exploratory Single-Arm Phase II Clinical Trail
Brief Title: Stereotactic Radiosurgery Combination With Anlotinib for Limited Brain Metastases With Perilesional Edema in NSCLC
Acronym: Rvision-001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Huashan Hospital (Other); Tianjin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rvision-001
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-10

CONDITIONS: Stereotactic Body Radiation Therapy
MeSH Terms: interventions — anlotinib; Angiogenesis Inhibitors; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRS Combination With Anlotinib (Experimental): Stereotactic Radiosurgery Combination With Anlotinib
  Interventions: Drug: Anlotinib; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Drug: Anlotinib — Anlotinib is a novel multi-target tyrosine Kinase inhibitor that inhibits VEGFR2/3, FGFR1-4, PDGFD α/β, c-Kit and Ret.
  Other Names: Antiangiogenic agents
Radiation: Stereotactic Radiosurgery — Stereotactic Radiosurgery as the initial treatment of non small cell lung cancer patients with limited brain metastases

SUMMARY:
The purpose of this study is to determine whether stereotactic radiosurgery combination with Anlotinib is safe, effective in the treatment of limited brain metastases with Perilesional edema in non-small cell lung cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether stereotactic radiosurgery combination with Anlotinib is safe, effective in the treatment of limited brain metastases with perilesional edema in non-small cell lung cancer. The sample size is 50. Patients start to take Anlotinib 1 week before the MRI-based simulation，12mg/d QD，day1~14, day22~36.Edema index will be used to evaluate the effectiveness of Anlotinib. The "Edema index (EI)" is calculated per the equation of "edema index= (peri-tumoral edema volume+ tumor volume)/tumor volume.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, signed informed consent.
2. Patients pathologically diagnosed as non-small cell lung cancer, with brain metastases and measurable lesions;
3. Patients aged between 18 -80 years; with expected survival time>3 months.
4. Patients with no more than 5 brain metastases
5. Patients with normal organ function within 7 days prior to treatment, the following criteria are met:

   a) blood routine examination criteria : i) hemoglobin (HB) ≥90g/L; ii) absolute neutrophil count (ANC) ≥1.5×10e9/L; iii) platelet (PLT) ≥80×10e9/L; b) biochemical tests meet the following criteria: i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; iii) serum creatinine (Cr) ≤1.5 ULN or creatinine clearance (CCr) ≥60mL/min;
6. Female patients should agree to use contraceptives during and within 6 months after the study.

Exclusion Criteria:

1. Patients who had previously used antiangiogenic agents within 1 month;
2. Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer);
3. Patient with lung squamous cell carcinoma that involved pulmonary hilar, or non-small cell lung cancer with hemoptysis;
4. Patients with cerebral infarction and cerebral hemorrhage;
5. Patients without perilesional edema；
6. Patients with more than grade 2 (NCI-CTCAE v4.0) acute toxicity reaction due to any previous treatment.
7. Patients with factors that affect oral medication (such as cannot swallow, chronic diarrhea and intestinal obstruction, etc.);
8. Patients with visceral dissemination or severe symptoms, which could cause death in short term;
9. Patients with any other severe and/or uncontrolled disease;
10. Patients who received a surgery, a biopsy or a significant traumatic injury within 1 month;
11. Patients with any signs or medical history of bleeding, unhealed wounds, ulcers or fractures, regardless of the severity;
12. Patients underwent artery or venous thrombotic events within 2 months, such as deep vein thrombosis and pulmonary embolism;
13. Patients with a history of psychotropic medicine abuse and cannot quit or have mental disorders;
14. Patients with disease which will severely endanger their security and could not complete this study, according to the judgement of researchers；
15. Patients who still can't tolerate SRS after anlotinib treatment, even after adding mannitol, and have to receive steroid treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-24 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
EI | 1 month
  Edema Index. The "Edema index (EI)" is calculated per the equation of "edema index= (peri-tumoral edema volume+ tumor volume)/tumor volume.

SECONDARY OUTCOMES:
PFS | 1 year
  Progression-free Survival
OS | 1 year
  Overall Survival
ORR | 3 months
  Objective Response Rate
DCR | 3 months
  Disease Control Rate
iORR | 3 months
  intracranial objective response rate
iPFS | 3 months
  intracranial progression-free survival
SRS rate | 1 month
  the rate of SRS after anlotinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hongqing Zhuang, doctor, Study Director — Peking University Third Hospital
Locations (1):
- Department of Radiation Oncology Cancer Center, Peking University Third Hospital 49# North Garden Rd.,Haidian Dist., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhuang H, Wang Y, Cheng C, Shi S. The efficacy of anlotinib instead of glucocorticoids for edema induced by brain metastases in NSCLC patients with anti-PD1/PDL-1 immunotherapy. Neuro Oncol. 2021 Jan 30;23(1):169-171. doi: 10.1093/neuonc/noaa236. No abstract available. PMID 33294918